CLINICAL TRIAL: NCT01199380
Title: Stage II Trial of Novel Behavioral Activation Intervention for Smoking Cessation
Brief Title: Behavioral Activation Intervention for Smoking Cessation in Smokers With Depressive Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Laura MacPherson, Dr. Laura MacPherson, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA018730; 5R01DA018730-07 (NIH)
Record Dates: First submitted 2010-09-03; First posted 2010-09-10 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Cigarette Smoking
Keywords: Smoking, Smoking Cessation
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation | interventions — Smoking Devices; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Treatment (ST) (Active Comparator): Participants will receive a standard, group smoking cessation treatment equated for contact time, based on the most recent clinical practice guideline for treating tobacco. Treatment will be delivered in 8, 60-minute group sessions over an 8-week period. Patients in ST will complete between group exercises and will also keep a weekly written journal throughout treatment elaborating on observations about the day's events, their thoughts, feelings, and insights about their reactions to these events. Participants will also receive 8 weeks of the transdermal nicotine patch.
  Interventions: Behavioral: Standard Treatment; Drug: Transdermal Nicotine Patch
- Behavioral Activation for Smoking (Experimental): Behavioral Activation Treatment for Smoking (BATS) includes standard smoking cessation strategies and identifying life areas, values, and daily activities to help manage mood. Participants will complete between group exercises and will also monitor and plan daily activities in line with their values. Treatment will be delivered in 8, 60-minute group sessions over an 8-week period. Participants will also receive 8 weeks of the transdermal nicotine patch.
  Interventions: Behavioral: Behavioral Activation Treatment for Smoking; Drug: Transdermal Nicotine Patch

INTERVENTIONS:
Behavioral: Standard Treatment — Participants will receive a standard, group smoking cessation treatment, based on the most recent clinical practice guideline for treating tobacco use from the U.S. Department of Health and Human Services. Treatment will be delivered in 8, 60-minute group sessions over an 8-week period. Patients in ST will also keep a weekly written journal throughout treatment elaborating on observations about the day's events, their thoughts, feelings, and insights about their reactions to these events as a means to equate for time spent on daily activity monitoring in the BATS condition.
  Other Names: ST
  Arms: Standard Treatment (ST)
Behavioral: Behavioral Activation Treatment for Smoking — BATS is focused on identifying life areas, values, and daily activities to help one live according to his or her values. Treatment will be delivered in 8, 60-minute group sessions over an 8-week period.
  Other Names: BATS
  Arms: Behavioral Activation for Smoking
Drug: Transdermal Nicotine Patch — 8 weeks of the Transdermal Nicotine Patch Nicoderm CQ at 24 hour doses of 21, 14, and 7 mg respectively depending on participant's initial level of nicotine use. Nicotine patch dose will decrease at 2 or 4 week increments also specific to the participant's initial nicotine level.
  Other Names: Nicoderm CQ

SUMMARY:
Depression related vulnerabilities are highly comorbid with smoking behavior and dramatically reduce cessation rates among both community and clinical samples. Previous research has examined the efficacy of cognitive-behavioral treatment for individuals with a history of major depressive disorder (MDD) in standard cessation treatment. A broader health impact can be achieved by targeting individuals with current elevated depressive symptoms to address their association with cessation failure. Thus the objective of the present proposal is to conduct a Stage II randomized controlled trial (RCT) comparing the behavioral activation intervention to standard treatment among a similar community sample of 200 adult smokers with elevated depressive symptoms. Participants will be followed over 52 weeks post-quit date and the larger sample size will allow for more complex analysis of cessation outcomes.

DETAILED DESCRIPTION:
This will be a Stage II randomized control trial to examine the efficacy of behavioral activation treatment for smoking (BATS) vs. standard smoking cessation treatment (ST). We will recruit 200 smokers with elevated depressive symptoms who will be randomized into one of two treatment groups. Treatment will be delivered in group format across both the BATS (n = 100) and ST condition (n = 100). All participants will receive 8 weeks of transdermal nicotine patch in addition to their assigned treatment group. We intend to compare the BA treatment for smoking (BATS) to a standard smoking cessation intervention (ST)on abstinence and relapse outcomes. In addition we will examine to what extent depressive symptoms and reward sensitivity prior to quit date will mediate the effects of BATS on improved smoking cessation outcomes relative to ST.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age
* A regular smoker for at least one year
* Currently smoking an average of at least 10 cigarettes per day
* Want to quit smoking
* Report current elevated depressive symptoms

Exclusion Criteria:

* Current Axis I disorder
* Psychoactive substance dependence (excluding nicotine dependence) within the past 6 months
* Current use of psychotropic medication or participation in any form of psychotherapy
* A history of significant medical condition (e.g., cardiovascular , neurological, gastrointestinal), pregnancy and/or breast feeding, or other systemic illness
* Current use of any pharmacotherapy for smoking cessation not provided by the researchers during the quit attempt

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura MacPherson, PhD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, College Park, College Park, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment (ST): Eight, 60-minute group sessions over an 8-week period. Participants will also receive 8 weeks of the transdermal nicotine patch.
  Eight weeks of transdermal nicotine patch, which will begin at the time of quitting smoking and will continue even after the treatment sessions have ended. Standard nicotine patch dosing will be used.
  Transdermal Nicotine Patch: 8 weeks of the Transdermal Nicotine Patch Nicoderm CQ at 24 hour doses of 21, 14, and 7 mg respectively depending on participant's initial level of nicotine use. Nicotine patch dose will decrease at 2 or 4 week increments also specific to the participant's initial nicotine level.
- Behavioral Activation for Smoking: Behavioral Activation Treatment for Smoking (BATS) includes standard smoking cessation strategies and identifying life areas, values, and daily activities to help manage mood. Eight, 60-minute group sessions over an 8-week period. Participants will also receive 8 weeks of the transdermal nicotine patch.
  Eight weeks of transdermal nicotine patch, which will begin at the time of quitting smoking and will continue even after the treatment sessions have ended. Standard nicotine patch dosing will be used.
  Transdermal Nicotine Patch: 8 weeks of the Transdermal Nicotine Patch Nicoderm CQ at 24 hour doses of 21, 14, and 7 mg respectively depending on participant's initial level of nicotine use. Nicotine patch dose will decrease at 2 or 4 week increments also specific to the participant's initial nicotine level.
Period: Overall Study
Arm/Group | Standard Treatment (ST) | Behavioral Activation for Smoking
Started | 88 | 96
Completed | 78 | 81
Not Completed | 10 | 15

BASELINE CHARACTERISTICS:
Population: Analysis population is not different from the assignment in Participant Flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment (ST) | Behavioral Activation for Smoking | Total
Number analyzed (Participants) | 88 | 96 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 87 | 96 | 183
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.25 (10.38) | 44.02 (12.47) | 44.61 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 82
  Male | 45 | 57 | 102
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 65 | 74 | 139
  White | 9 | 12 | 21
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 88 | 96 | 184

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Smoking-Abstinent for 7 Days, 52 Weeks Post Quit Date
Description: 7 days of smoking abstinence confirmed biochemically at 52 week post quit attempt
Time Frame: 52 weeks post quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment (ST) | Behavioral Activation for Smoking
Number analyzed (Participants) | 88 | 96
Participants | 26 | 19

ADVERSE EVENTS:
Time Frame: 3 years, 8 months
Description: Definition of adverse event and/or serious adverse event does not differ from clinicaltrials.gov definitions.
Groups:
- Standard Treatment (ST): One 60-minute individual session Seven 2-hour group sessions Two individual brief telephone contacts over an eight-week period. Eight weeks of transdermal nicotine patch, which will begin at the time of quitting smoking and will continue even after the treatment sessions have ended. Standard nicotine patch dosing will be used.
  Transdermal Nicotine: Participants will use the full strength 21mg. patch for 4 weeks, will taper to the 14 mg. patch for the next 2 weeks, and then to the 7 mg. patch for the remaining 2 weeks of treatment.
Arm/Group | Standard Treatment (ST) | Behavioral Activation for Smoking
All-Cause Mortality (participants affected / at risk) | 2/88 | 0/96
Serious Adverse Events (participants affected / at risk) | 2/88 | 1/96
Other Adverse Events (participants affected / at risk) | 0/88 | 0/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment (ST) (N=88) | Behavioral Activation for Smoking (N=96)
Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Throat cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No